CLINICAL TRIAL: NCT03572348
Title: VeSpAR: A Randomized Controlled Trial Comparing Vessel-Sparing Anastomotic Repair and Transecting Anastomotic Repair in Isolated Short Bulbar Urethral Strictures
Brief Title: VeSpAR: Comparing Vessel-Sparing Anastomotic Repair and Transecting Anastomotic Repair in Isolated Short Bulbar Strictures.
Acronym: VeSpAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC-03662
Record Dates: First submitted 2018-06-05; First posted 2018-06-28 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Urethral Stricture; Surgery; Urologic Diseases
Keywords: urethral stricture; urethroplasty; bulbar urethra; reconstructive surgery; lower urinary tract symptoms; erectile function
MeSH Terms: conditions — Urethral Stricture; Urologic Diseases; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, multicentric, single-blinded, randomized, controlled, non-inferiority, phase II trial
Who Masked: Participant
Masking Description: Patients will be randomized using software in a 1:1 ratio in either the vessel-sparing group or the transecting group. Randomisation will be stratified per participating center and single blinded; double blindation is impossible as the surgeon has to know which technique to perform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transecting anastomotic repair (tAR) (Active Comparator): Classic technique, which involves full thickness transection of the corpus spongiosum and the embedded urethral blood supply.
  Interventions: Procedure: Transecting anastomotic repair (tAR)
- Vessel-sparing anastomotic repair (vsAR) (Active Comparator): Alternative technique, leaving the bulbar arteries intact, only transecting and excising the narrow segment of the urethra and the surrounding spongiofibrosis.
  Interventions: Procedure: Vessel-sparing anastomotic repair (vsAR)

INTERVENTIONS:
Procedure: Transecting anastomotic repair (tAR) — Classic technique, which involves full thickness transection of the corpus spongiosum and the embedded urethral blood supply.
  Arms: Transecting anastomotic repair (tAR)
Procedure: Vessel-sparing anastomotic repair (vsAR) — Alternative technique, leaving the bulbar arteries intact, only transecting and excising the narrow segment of the urethra and the surrounding spongiofibrosis.
  Arms: Vessel-sparing anastomotic repair (vsAR)

SUMMARY:
The investigators want to verify whether the surgical outcome of vessel-sparing anastomotic repair in isolated short bulbar urethral strictures is not inferior to the surgical outcome of transecting anastomotic repair. Furthermore, the investigators compare the functional outcome of both techniques verifying if there is less erectile dysfunction after vessel-sparing anastomotic repair than after transecting anastomotic repair.

DETAILED DESCRIPTION:
A randomized controlled trial comparing vessel-sparing anastomotic repair (vsAR) and transecting anastomotic repair (tAR) in isolated short bulbar urethral strictures (maximum 3 centimeter) for both surgical and functional outcome, to demonstrate that vsAR is not inferior to tAR regarding the surgical outcome, and to demonstrate a benefit for vsAR over tAR regarding postoperative erectile function.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signed written informed consent (according to the rules of Good Clinical Practice and national regulations)
* Male
* Age >= 18 years
* Fit for operation, based on the surgeon's expert opinion
* Isolated short (=< 3cm) bulbar urethral stricture confirmed by preoperative retrograde urethrography (RUG), voiding cysto-urethrography (VCUG), cystoscopy, ultrasonography or a combination of investigations
* Unique urethral stricture
* Urethral stricture =< 3 cm
* Urethral stricture at the bulbar segment
* Patient declares that it will be possible for him to attend the follow-up consultation

Exclusion Criteria:

* Absence of signed written informed consent
* Age <18 years
* Female patients
* Transgender patients
* Patients unfit for operation
* Concomitant urethral strictures at other urethral locations (penile urethra, membranous urethra, prostatic urethra, bladder neck)
* Urethral strictures exceeding 3 cm
* A unique urethral stricture at other urethral locations (penile urethra, membranous urethra, prostatic urethra, bladder neck)
* Lichen Sclerosus related strictures
* Strictures after failed hypospadias repair
* Patients with neurogenic bladder
* Shift of technique to augmented urethroplasty due to any circumstance
* History of pelvic radiation therapy
* Active treatment to enhance erectile function (such as PDE5-inhibitors and intracavernous injections) at the moment of prescreening for inclusion in this trial
* Any condition or situation, which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study
* Patient declares that it will be impossible for him to attend the follow-up consultations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
FFS at 24 months | 24 months
  Failure-free survival at 24 months. Surgical failure is defined as urethroscopic evidence of stricture recurrence, impossible to pass with a 16Fr silicone urethral catheter, independent of whether the stricture is treated or not.

SECONDARY OUTCOMES:
FFS at 3 and 12 months | 3 and 12 months
  Failure-free survival at 3 and 12 months. Surgical failure is defined as urethroscopic evidence of stricture recurrence, impossible to pass with a 16Fr silicone urethral catheter, independent of whether the stricture is treated or not.
Erectile function | 3, 12, and 24 months
  Erectile function score assessed by the International Index of Erectile Function (IIEF-5) questionnaire
Ejaculatory function | 3, 12, and 24 months
  Ejaculatory function score assessed by the Male Sexual Health Questionnaire - Ejaculatory Dysfunction short form (MSHQ-EjD short form)
Voiding function | 3, 12, and 24 months
  Lower Urinary Tract symptoms assessed by the Peeling's voiding picture.
Lower Urinary Tract symptoms | 3, 12, and 24 months
  Lower Urinary Tract symptoms assessed by the International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms module (ICIQ-MLUTS)
Urinary incontinence | 3, 12, and 24 months
  Urinary incontinence assessed by the International Consultation on Incontinence Questionnaire - Urinary Incontinence short form (ICIQ-UI)
Maximum flow rate | 3, 12, and 24 months
  Qmax assessed using uroflowmetry
Residual urinary volumes | 3, 12, and 24 months
  Residual urinary volumes examined by suprapubic ultrasonic measurement after voiding
Quality of life (EQ-5D-3L) | 3, 12, and 24 months
  QoL scored by the EQ-5D-3L questionnaire
Quality of life (EQ-VAS) | 3, 12, and 24 months
  QoL scored by the EQ visual analogue scale (EQ-VAS)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - Department of Urology, SUNY Upstate Medical University, Syracuse, New York
  - Department of Urology, Eastern Virginia Medical School, Norfolk, Virginia
- Argentina (2):
  - Department of Urology, Centro de Educación Médica e Investigaciones Clínicas, Buenos Aires
  - Department of Urology, Hospital Italiano de Buenos Aires, Buenos Aires
- Belgium (2):
  - Dept. of Urology, Ghent University Hospital, Ghent
  - Dept. of Urology, University Hospital Leuven, Leuven
- Department of Urology, Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, China
- Mexico (2):
  - Centro de Uretra Las Alamedas, Mexico City
  - Department of Urology, Hospital San José Tecnológico de Monterrey, Universidad de Monterrey, Monterrey
- Department of Urology, Hospital de Santa María, Universidad de Lisboa, Lisbon, Portugal
- Spain (2):
  - Department of Urology, Departamento Clínico, Facultad de Ciencias Biomédicas, Universidad Europea de Madrid, Hospital Universitario de Getafe, Madrid
  - Dept. of Urology, Hospital Univ. de Valdecilla, Santander
- Department of Urology, University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Latini JM, McAninch JW, Brandes SB, Chung JY, Rosenstein D. SIU/ICUD Consultation On Urethral Strictures: Epidemiology, etiology, anatomy, and nomenclature of urethral stenoses, strictures, and pelvic fracture urethral disruption injuries. Urology. 2014 Mar;83(3 Suppl):S1-7. doi: 10.1016/j.urology.2013.09.009. Epub 2013 Nov 8. PMID 24210733
- [Background] Palminteri E, Berdondini E, Verze P, De Nunzio C, Vitarelli A, Carmignani L. Contemporary urethral stricture characteristics in the developed world. Urology. 2013 Jan;81(1):191-6. doi: 10.1016/j.urology.2012.08.062. Epub 2012 Nov 13. PMID 23153951
- [Background] Morey AF, Watkin N, Shenfeld O, Eltahawy E, Giudice C. SIU/ICUD Consultation on Urethral Strictures: Anterior urethra--primary anastomosis. Urology. 2014 Mar;83(3 Suppl):S23-6. doi: 10.1016/j.urology.2013.11.007. Epub 2013 Dec 27. PMID 24373726
- [Background] Jordan GH, Eltahawy EA, Virasoro R. The technique of vessel sparing excision and primary anastomosis for proximal bulbous urethral reconstruction. J Urol. 2007 May;177(5):1799-802. doi: 10.1016/j.juro.2007.01.036. PMID 17437823
- [Background] Gur U, Jordan GH. Vessel-sparing excision and primary anastomosis (for proximal bulbar urethral strictures). BJU Int. 2008 May;101(9):1183-95. doi: 10.1111/j.1464-410X.2008.07619.x. No abstract available. PMID 18399836
- [Background] Lumen N, Poelaert F, Oosterlinck W, Lambert E, Decaestecker K, Tailly T, Hoebeke P, Spinoit AF. Nontransecting Anastomotic Repair in Urethral Reconstruction: Surgical and Functional Outcomes. J Urol. 2016 Dec;196(6):1679-1684. doi: 10.1016/j.juro.2016.06.016. Epub 2016 Jun 12. PMID 27307398
- [Background] Andrich DE, Mundy AR. Non-transecting anastomotic bulbar urethroplasty: a preliminary report. BJU Int. 2012 Apr;109(7):1090-4. doi: 10.1111/j.1464-410X.2011.10508.x. Epub 2011 Sep 20. PMID 21933325
- [Background] Virasoro R, Zuckerman JM, McCammon KA, DeLong JM, Tonkin JB, Capiel L, Rovegno AR, Favre G, Giudice CR, Eltahawy EA, Gur U, Jordan GH. International multi-institutional experience with the vessel-sparing technique to reconstruct the proximal bulbar urethra: mid-term results. World J Urol. 2015 Dec;33(12):2153-7. doi: 10.1007/s00345-015-1512-9. Epub 2015 Feb 18. PMID 25690318
- [Background] Bugeja S, Andrich DE, Mundy AR. Non-transecting bulbar urethroplasty. Transl Androl Urol. 2015 Feb;4(1):41-50. doi: 10.3978/j.issn.2223-4683.2015.01.07. PMID 26816808
- [Background] Anderson KM, Blakely SA, O'Donnell CI, Nikolavsky D, Flynn BJ. Primary non-transecting bulbar urethroplasty long-term success rates are similar to transecting urethroplasty. Int Urol Nephrol. 2017 Jan;49(1):83-88. doi: 10.1007/s11255-016-1454-1. Epub 2016 Nov 14. PMID 27844407
- [Background] Le W, Li C, Zhang J, Wu D, Liu B. Preliminary clinical study on non-transecting anastomotic bulbomembranous urethroplasty. Front Med. 2017 Jun;11(2):277-283. doi: 10.1007/s11684-017-0515-x. Epub 2017 Apr 22. PMID 28432540
- [Background] Andrich DE, Dunglison N, Greenwell TJ, Mundy AR. The long-term results of urethroplasty. J Urol. 2003 Jul;170(1):90-2. doi: 10.1097/01.ju.0000069820.81726.00. PMID 12796652
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Utomo E, Blok BF, Pastoor H, Bangma CH, Korfage IJ. The measurement properties of the five-item International Index of Erectile Function (IIEF-5): a Dutch validation study. Andrology. 2015 Nov;3(6):1154-9. doi: 10.1111/andr.12112. Epub 2015 Oct 9. PMID 26453539
- [Background] Verla W, Waterloos M, Lumen N. Urethroplasty and Quality of Life: Psychometric Validation of a Dutch Version of the Urethral Stricture Surgery Patient Reported Outcome Measures. Urol Int. 2017;99(4):460-466. doi: 10.1159/000479189. Epub 2017 Aug 30. PMID 28850951
- [Background] Lesaffre E. Superiority, equivalence, and non-inferiority trials. Bull NYU Hosp Jt Dis. 2008;66(2):150-4. PMID 18537788
- [Background] Rubinstein LV, Korn EL, Freidlin B, Hunsberger S, Ivy SP, Smith MA. Design issues of randomized phase II trials and a proposal for phase II screening trials. J Clin Oncol. 2005 Oct 1;23(28):7199-206. doi: 10.1200/JCO.2005.01.149. PMID 16192604
- [Derived] Verla W, Waterloos M, Waterschoot M, Van Parys B, Spinoit AF, Lumen N. VeSpAR trial: a randomized controlled trial comparing vessel-sparing anastomotic repair and transecting anastomotic repair in isolated short bulbar urethral strictures. Trials. 2020 Sep 11;21(1):782. doi: 10.1186/s13063-020-04712-5. PMID 32917251